CLINICAL TRIAL: NCT05880017
Title: Modified Versus Conventional Thoracolumbar Interfascial Plane Block for Perioperative Analgesia in Lumber Spine Surgery. A Randomized Controlled Study.
Brief Title: Thoracolumbar Interfascial Plane Block in Lumber Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Diaaeldein Mahmoud Haiba, Lecturer of Anesthesia, ICU and Pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 167/2022
Record Dates: First submitted 2023-05-05; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Post Operative Pain Management
Keywords: Thoracolumber; Interfascial plane; Lumber discectomy
MeSH Terms: interventions — Dental Occlusion; Morphine; Control Groups; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Prospective , randomized controlled, comparative study.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modified Group (Active Comparator): A total of 20 patients undergoing lumber spine surgery receiving modified ultrasound guided thoracolumbar interfascial plane (TLIP) block.
  Interventions: Procedure: Modified ultrasound guided thoracolumbar interfascial plane (TLIP) block.; Drug: Bupivacain
- Conventional Group (Active Comparator): A total of 20 patients undergoing lumber spine surgery receiving conventional ultrasound guided thoracolumbar interfascial plane (TLIP) block.
  Interventions: Procedure: Conventional ultrasound guided thoracolumbar interfascial plane (TLIP) block.; Drug: Bupivacain
- Morphine Group (Active Comparator): A total of 20 patients undergoing lumber spine surgery receiving morphine for peritoperative analgesia (control group).
  Interventions: Drug: Morphine for peritoperative analgesia (control group).

INTERVENTIONS:
Procedure: Modified ultrasound guided thoracolumbar interfascial plane (TLIP) block. — Patients will be placed in a prone position; modified ultrasound guided TLIP block will be performed using a SonoSite 2-5 MHZ Curved array (C60X) transducer. The transducer will be positioned in a transverse midline position at the level of the L3 vertebra. After the identification of the spinous process and interspinous muscles, the probe will be moved laterally to identify longissimus (LG) and intercostalis muscles. After identifying the muscles and decontamination of the skin, the modified TLIP block will be performed under real-time ultrasound guidance using an insulated 90-mm 22G echogenic needle which will be inserted at a 15ºangle from the skin in-plane in a medial to lateral direction injecting the anesthetic locally between the longissimus and intercostalis muscles, which are easy to define using ultrasonography. After negative aspiration, injection will be in each side bilaterally in the interface between the LG and intercostalis muscles.
  Arms: Modified Group
Procedure: Conventional ultrasound guided thoracolumbar interfascial plane (TLIP) block. — Patients will be placed in a prone position; conventional ultrasound guided TLIP block will be performed using a SonoSite 2-5 MHZ Curved array (C60X) transducer. The transducer will be positioned in a transverse midline position at the level of the L3 vertebra. After the identification of the spinous process and interspinous muscles, the probe will be moved laterally to identify the multifidus (MF) and longissimus (LG) muscles. After identifying the muscles and decontamination of the skin, the TLIP block will be performed under real-time ultrasound guidance using an insulated 90-mm 22G echogenic needle which will be inserted at a 30ºangle from the skin in-plane lateral to the medial direction through the belly of the LG toward the MF muscle. After negative aspiration, injection will be done in each side bilaterally in the interface between the MF and LG muscles.
  Arms: Conventional Group
Drug: Morphine for peritoperative analgesia (control group). — Morphine based analgesia, after emergence they will receive 5mg morphine IV as a start and the rest of the first 24 hours they will receive incremental dose of intravenous morphine according to pain score.
  Arms: Morphine Group
Drug: Bupivacain — As a local anesthetic will be injected in modified and conventional groups 20ml in each side.
  Arms: Conventional Group; Modified Group

SUMMARY:
The goal of this clinical trial is to compare modified versus conventional thoracolumbar interfascial plane block for perioperative analgesia in lumber spine surgery.

The main question it aims to answer is:

• Whether modified thoracolumbar interfascial plane block is as effective as the conventional block for perioperative analgesia in lumber spine surgery.

60 patients were enrolled in the study, divided by simple random sampling into 3 groups.

DETAILED DESCRIPTION:
Spinal surgeries are usually associated with marked postoperative pain that classically takes 3 days to recede.

Adequate perioperative pain control is significant for patients to encourage early mobilization and reduce postoperative adverse events. Discectomy, laminectomy, and spinal fixation are the most frequently performed spinal surgical procedures. Extensive dissection of tissues, ligaments, and bones is often performed during spinal surgeries, resulting in a significant degree of postoperative severe pain. Adequate pain management in these patients is challenging because most of them have already received ordinary analgesics and/or opioids to ameliorate preexistent chronic back pain. Pain following spine surgery can result from mechanical irritation, nerve compression, or postoperative inflammatory processes. It can be generated from different structures such as vertebrae, discs, ligaments, muscles, dural sleeves, and capsules of the facet joint. Innervation of these pain generators is from the dorsal rami of spinal nerves. Opioids are considered the standard method of analgesia and are commonly used as effective analgesics for the management of severe pain disorders. However, their widespread use is restricted because of their side effects such as nausea, vomiting, and respiratory distress, and acquired tolerance. Preemptive multimodal analgesic regimens that rely on the synergistic action of nonopioid agents given in lower doses have been used to improve postoperative pain management and reduce opioid consumption. Protocols for reducing pain after lumbar surgery recommend the use of regional anesthesia techniques to reduce opioid analgesic use to the minimum. Interfascial plane blocks have the potential to provide extended postoperative analgesia and to reduce opioid consumption and neuraxial-related motor block to a minimum. The use of thoracolumbar interfascial plane block TLIP block was first reported in 2015 by Hand et al. wherein they did a volunteer-based study and demarcated the area of sensory analgesia. Thereafter, Ueshima et al. reported two cases of spinal surgeries where TLIP block was administered. TLIP blocks the sensory component of the dorsal rami of the thoracolumbar nerves. These nerves emerge mainly through the interface between the multifidus (MF) and longissimus (LG) muscles. Blocking these nerves provides good analgesia after spine surgeries. TLIP modification where we inject the anaesthetics between the longissimus and iliocostalis muscles after having advanced the needles at a 15 angle in a medial to lateral direction. This modified method has several advantages. 1.Advancing the needle from a medial to lateral direction eliminates the risk of possible inadvertent neuraxial injection. 2.Injecting between the iliocostalis and longissimus muscles results in a dermatomal area of analgesia similar to that obtained with an injection made between the multifidus and longissimus muscles. Both conventional and modified techniques are assumed to be effective and safe.

The primary outcome measure is postoperative pain intensity expressed as A numerical rating scale (NRS) score at time zero (time of extubation), time 1 ( time of delivery to PACU), every 2 hours during the first 6 hours then every 6 hours during the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes admitted to the OR of Ain Shams University Hospitals for lumber disc surgery.
* Age 18 to 70 year old.
* ASA classification I and II.

Exclusion Criteria:

* Age <18 or >70 years.
* Declining to give written informed consent.
* History of allergy to the medications used in the study.
* Psychiatric disorder.
* ASA classification III-V.
* Patients with cerebrovascular accidents.
* Neuromuscular disorders, spine abnormalities.
* Spinal cord or head injuries.
* CNS tumours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain intensity expressed as A numerical rating scale (NRS) score at time zero (time of extubation). | Time 0 (Time of Extubation)
  The numerical rating scale consists of a numeric version of the visual analogue scale. The most common form of the NRS is a horizontal line with an eleven point numeric range.
  The numerical rating scale requires the patient to rate their pain on a defined scale. Numerical rating scale (NRS) is the simplest and most commonly used scale. The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."

SECONDARY OUTCOMES:
Pain intensity expressed as A numerical rating scale (NRS) score at time 1 (time of delivery to Post Anesthesia Care Unit PACU). | Time 1 (30 minutes after extubation in the Post Anesthesia Care Unit (PACU).
  The numerical rating scale consists of a numeric version of the visual analogue scale. The most common form of the NRS is a horizontal line with an eleven point numeric range.
  The numerical rating scale requires the patient to rate their pain on a defined scale. Numerical rating scale (NRS) is the simplest and most commonly used scale. The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."
Pain intensity expressed as A numerical rating scale (NRS) score at time 6 (6 hours postoperative). | Time 6 (6 hours postoperative)
  The numerical rating scale consists of a numeric version of the visual analogue scale. The most common form of the NRS is a horizontal line with an eleven point numeric range.
  The numerical rating scale requires the patient to rate their pain on a defined scale. Numerical rating scale (NRS) is the simplest and most commonly used scale. The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."
Pain intensity expressed as A numerical rating scale (NRS) score at time 24 (24 hours postoperative). | Time 24 (24 hours postoperative)
  The numerical rating scale consists of a numeric version of the visual analogue scale. The most common form of the NRS is a horizontal line with an eleven point numeric range.
  The numerical rating scale requires the patient to rate their pain on a defined scale. Numerical rating scale (NRS) is the simplest and most commonly used scale. The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."
Early ambulation. | Time of ambulation during first 24 hours postoperative
  Time of starting ambulation postoperative
Time of first rescue analgesic. | During First 24 hours postoperative.
  As-needed dose of opioid (morphine) to provide relief of first breakthrough pain.
Total dose of Postoperative morphine consumption during first 24 hours. | During first 24 hours.
  Dose of morphine in milligram

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university hospitals, Cairo, Al Abbassia, Egypt